CLINICAL TRIAL: NCT07399171
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2a Study to Evaluate the Effect of HT-4253 for the Prevention of Alzheimer's Disease in APOE4 Carriers
Brief Title: Study to Evaluate the Effect of HT-4253 for the Prevention of Alzheimer's Disease in APOE4 Carriers
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Halia Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HT-4253-APOE-002
Record Dates: First submitted 2025-12-24; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Alzheimers Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Arm HT-4253 (Active Comparator): Arm HT-4253:
  HT-4253 (300 mg): dosed once a day, orally (PO QD)
  Interventions: Drug: HT-4253
- Study Arm Placebo (Placebo Comparator): Arm Placebo:
  Placebo: Dosed once a day, orally (PO QD). Participants in this group will switch over to active treatment at week 24.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: HT-4253 — It is anticipated that 112 participants will be randomized to receive HT-4253 (56 in each study arm).
  Arms: Study Arm HT-4253
Other: Placebo — It is anticipated that 112 participants will be randomized to receive placebo (56 in each study arm).
  Arms: Study Arm Placebo

SUMMARY:
Primary Objectives:

To demonstrate that HT-4253 improves the amyloid risk profile by transitioning biomarker-positive APOE4 carriers from a positive, high risk APS2 score to a negative, low risk APS2 score.

Secondary Objectives:

* To assess the effects of HT-4253 on tau related blood biomarker progression over the study period.
* To assess the effects of HT-4253 on amyloid related blood biomarker progression over the study period.
* To assess the safety and tolerability of HT-4253 in the UAE population.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be 50-75 years of age, without previous AD diagnosis at the time of signing the informed consent.
2. Capable of giving signed informed consent.
3. Body mass index (BMI) between 18 and 32 kg/m2.
4. A positive amyloid probability score from PrecivityAD2™ test (≥ 47.5).
5. APOE4 carrier: homozygous (APOE4/APOE4) or heterozygous (APOE3/APOE4), confirmed using the Precivity-ApoE™ test.
6. Must be ambulatory.
7. Must be in good health, as determined by the PI, without clinically significant medical history.
8. Normal physical examination, 12-lead ECG, and vital signs, as determined by the PI.
9. Females must meet one of the following:

   * Postmenopausal
   * Surgically sterile
10. Male participants who are sexually active with a woman of childbearing potential must agree to use a double contraception during the study and for 30 days after the last dose of HT-4253.
11. Female participants must have a negative serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) at screening.
12. Able to comply with the study procedures in the view of the PI.

Exclusion Criteria:

1. Any medical or neurological condition that in the opinion of the PI may be supportive of dementia.
2. A history of subjective memory decline with gradual onset and slow progression over the 6 months prior to Screening.
3. Previous or current diagnosis of AD or mild cognitive decline: MoCA < 26.
4. Any clinically significant CNS, cardiac, pulmonary, renal, gastrointestinal, endocrinological, respiratory, or metabolic conditions (or history), or other pathological or physiological conditions, that might interfere with the study results in the PI's opinion.
5. Any condition which, in the PI's opinion, puts the participant at significant risk, could confound the study results, or may interfere significantly with the participant's participation in the study.
6. History of clinically significant unstable psychiatric illness at the PI's discretion (e.g., uncontrolled major depression, uncontrolled schizophrenia, uncontrolled bipolar affective disorder) Note: Well-controlled and stable major depressive disorder or anxiety is permitted.
7. Prior treatment with an investigational LRRK2 inhibitor or any investigational AD therapy within the 6 months prior to Screening.
8. Concomitant use of prescription medications primarily indicated for psychiatric disorders or neurodegenerative disease (e.g., antipsychotics, mood stabilizers, investigational agents) within 30 days prior to first dose of study drug (Study Day 1).
9. Transient ischemic attack or stroke or any unexplained loss of consciousness (e.g., fainting without a diagnosis) within 1 year prior to Screening.
10. Known cerebral or systemic vasculopathy.
11. History of seizure or convulsion within 3 years prior to Screening or progressive neurologic disease (Parkinson's with dementia, epilepsy with breakthrough seizures, normal pressure hydrocephalus, multiple sclerosis with recent relapse).
12. Have donated blood or had loss of blood of more than a single unit of blood within 8 weeks before Screening or intend to donate blood during the course of the study.
13. Poorly controlled diabetes mellitus, as defined by having dosage adjustment of diabetic medication within 3 months prior to first dose of study drug (Study Day 1).
14. History of unstable angina, myocardial infarction, and/or chronic heart failure.
15. Chronic, uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥ 95 mmHg).
16. Vaccinations within 10 days prior to Screening.
17. Use of any medications, including prescription, over the counter (OTC) medications, vitamins, herbal preparations, and supplements, that, in the opinion of the PI, may put the participant at higher risk for AEs, or impair the participant's ability to complete study procedures.
18. Use of other investigational drugs at the time of Screening or within 30 days or 5 half-lives prior to signing of the ICF, whichever is longer, or longer if required by local regulations.
19. History of heavy smoking (i.e., more than 10 cigarettes a day or the tobacco/nicotine equivalent) within 3 months of Screening or refuse to abstain from tobacco or nicotine-containing products throughout the duration of the study.
20. History of, or current substance use disorder, including heavy alcohol use.
21. Pregnant or breastfeeding.
22. Presence of any laboratory abnormalities at Screening.
23. Prolonged QT interval exclusions for QTcF >450 ms for males and >470 ms for females Note: Entry of any participant with an abnormal ECG must be approved and documented by signature of the PI or a medically qualified sub-investigator.
24. Impaired renal function with estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2026-04-03 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 48 weeks
  To evaluate that HT-4253 improves the amyloid risk profile by transitioning biomarker-positive APOE4 carriers from a positive, high risk APS2 score to a negative, lower risk APS2 score
Primary Endpoint | Week 48
  Proportion of participants demonstrating improvement in amyloid risk profile, as defined by movement from high risk APS2 category (≥ 47.5) at baseline to a lower APS2 category (< 47.5) at week 48, as measured by C2N Diagnostics' PrecivityAD2™ test*
Primary Endpoint | Week 48
  *C2N PrecivityAD2™ Amyloid Probability Score 2 (APS2) Categories:
  •Low Risk (< 47.5): Low likelihood of amyloid plaques in the brain, consistent with a negative amyloid Positron Emission Tomography (PET) scan
Primary Endpoint | Week 48
  • High Risk (≥ 47.5): A score within this range suggests that the participant is likely to have amyloid plaques, requiring further diagnostic evaluation

SECONDARY OUTCOMES:
Secondary Objectives | 12, 24, 36, 48 weeks
  Secondary Objectives:
  To evaluate the effects of HT-4253 on tau related blood biomarker progression over the study period
Secondary Endpoints | 12, 24, 36, 48 weeks
  •Change in slope of p-tau217 over 48 weeks.
Secondary Endpoints | 12, 24, 36, 48 weeks
  •Change from baseline in plasma p-tau217 at weeks 12, 24, 36, 48.
Secondary Endpoints | 12, 24, 36, 48 weeks
  •Change from baseline in plasma p-tau181 at week 12, 24, 36, 48.
Secondary Objectives | 12, 24, 36, 48 weeks
  To evaluate the effects of HT-4253 on amyloid related blood biomarker progression over the study period.
Secondary Endpoints | 12, 24, 36, 48 Weeks
  • Change from baseline in plasma Aβ42 at weeks 12, 24, 36, 48.
Secondary Endpoints | 12, 24, 36, 48 Weeks
  • Change from baseline in plasma Aβ40 at weeks 12, 24, 36, 48.
Secondary Endpoints | 12, 24, 36, 48 Weeks
  • Change from baseline in plasma Aβ42/ Aβ40 ratio at weeks 12, 24, 36, 48.
Secondary Objectives | 12, 24, 36, 48 weeks
  To evaluate the safety and tolerability of HT-4253 in the UAE population.
Secondary Endpoints | 12, 24, 36, 48 weeks
  • Incidence and severity of treatment emergent adverse events (TEAEs).
Secondary Endpoints | 12, 24, 36, 48 weeks
  • Incidence of serious adverse events (SAEs).
Secondary Endpoints | 12, 24, 36, 48 weeks
  • Incidence and severity of treatment-related adverse events (TRAEs)
Secondary Endpoints | 12, 24, 36, 48 weeks
  • Incidence of discontinuations due to adverse events (AEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Abu Dhabi, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No